CLINICAL TRIAL: NCT06169878
Title: Evaluation of the Efficiency of the Adjustable Lower Extremity Abduction Apparatus After Total Hip Replacement Surgery
Brief Title: Efficiency of the Adjustable Lower Extremity Abduction Apparatus After Total Hip Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Tuğba Türkkan, Nurse, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BAHCESEHİRU-TTÜRKKAN-005
Record Dates: First submitted 2023-11-25; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Total Hip Replacement
Keywords: Total Hip Replacement; Adjustable Lower Extremity Abduction Apparatus; Gait; Dislocation
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): After total hip hip replacement surgery, the abduction apparatus, which provides abduction in the lower extremities and can be adjusted according to the height and weight of the patients, was used while lying and walking.
  Interventions: Device: Adjustable lower limb abduction apparatus
- control group (No Intervention): Pillows routinely used in the field were used to ensure abduction after total hip replacement surgery.

INTERVENTIONS:
Device: Adjustable lower limb abduction apparatus — To ensure abduction in the lower extremities after total hip replacement surgery, a specially adjustable apparatus developed according to the height and weight of each individual was used.
  This developed product was used by patients while they were lying down and walking.
  Arms: experimental group

SUMMARY:
This study was conducted to evaluate the effect of the adjustable lower extremity abduction apparatus developed after total hip arthroplasty (TKP) surgeries on preventing dislocation and walking.The study is of randomized controlled type. It was held on the inpatient floor of a Training and Research Hospital in Istanbul, between November 2021 and October 16, 2023, with patients undergoing femoral neck fracture surgery.

All patients who were admitted to this clinic for surgical intervention constituted the population of the study. In the research, 30 patients between the ages of 50-80 were included in the experimental group in which the "Adjustable lower extremity abduction apparatus" developed within the scope of the thesis was used, and 30 patients in which this apparatus was not used were included in the control group. As data collection tools in the study, "Patient Introduction Form", "Standardized Mini Mental State Test", "Patient Mobility Scale", "Modified Barthel Activities of Daily Living Index", "Apparatus Quality and Comfort Assessment Form" " and "Harris Hip Score Form" were used. Data were evaluated using IBM SPPS 27.0 statistical package program.

DETAILED DESCRIPTION:
This study aimed to evaluate the effect of an adjustable lower extremity abduction apparatus on the prevention of dislocation, activities of daily life and gait after total hip replacement (THR). The study was a randomised controlled trial. It was conducted on the inpatient floor of a Training and Research Hospital in Istanbul between November 2021 and 16 October 2023 with patients who had femoral neck fracture surgery. All patients admitted to this clinic for surgical intervention constituted the population of the study. In the study, 30 patients aged 50-80 years were included in the intervention group using the adjustable lower extremity abduction apparatus developed within the scope of the thesis, and 30 patients using the pillow in routine practice were included in the control group. Patient Introduction Form, Standardized Mini-Mental State Test, Patient Mobility Scale, Modified Barthel Activities of Daily Living Index, Apparatus Quality and Comfort Assessment Form, and Harris Hip Score Form were used as data collection tools. Data were analysed using the IBM SPPS 27.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 35 kg/m²,
* Femoral neck fractures,
* Patients who underwent hip arthroplasty due to femoral neck fracture,
* Those between the ages of 50-80,
* Those who do not have communication barriers,
* Patients without mental and cognitive dysfunction (Standardized mini mental state assessment test score between 24-30),
* Patients who agreed to participate in the study were included in the study

Exclusion Criteria:

* Patients who underwent hip arthroplasty due to coxarthrosis in advanced age,
* Those who use equipment as a walking aid before surgery,
* Those whose leg length difference is 3 cm or more,
* Patients who were operated on on one side and those with pathology in their other hips,
* Among patients who were operated on bilaterally, those with one side elevated,
* Those who have additional neuromuscular diseases (Multiple sclerosis, myasthenia gravis etc.),
* Those who have cancer,
* Those who are planned to undergo total hip replacement surgery due to pathological fractures,
* Those with diabetic feet that may prevent walking,
* Those who have previously had total hip replacement surgery,
* Other factors that cause dislocation development (Posterior surgical approach, incorrect position of one or both components, attachment of the femur to the pelvis or residual osteophytes, wedging of the neck of the femoral component to the edge of the acetabular component, insufficient soft tissue tension, size of the incision, inadequate or weak abductor muscle group , major trochanter avulsion or pseudoarthrosis, incompatibility and excessive positioning in the perioperative period, patient education, personal circumstances of the surgeon and the patient) were not included in the scope of the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
dislocation | 4-6 weeks
  Dislocation was determined by the patients electronic records and classified as "yes" or "no" depend on the presence or absence of the status
Activities of daily living | 4-6 weeks
  Daily living activities was assessed by using modified barthel actirivites of daily living index The modified Barthel Activities of Daily Living Index (MBGADLI) was developed by Barthel and Mahoney in 1965. Küçükdeveci et al. conducted a validity and reliability study of the index for the Turkish society with neurological patients in 2000. The Modified Barthel Index is an unbiased, easy-to-apply, understandable and causal relationship scale. The scores of the Modified Barthel Index for Activities of Daily Living range from 0 to 100. Higher scores indicate a greater level of independence.
Gait | 4-6 weeks
  Harris Hip Score was used to assess the patients gait Harris Hip Score (HHS): The Harris Hip Score, developed by W.H. Harris in 1969, evaluates patients who have undergone total hip replacement. Çelik et al. (2014) reported that the Turkish version of the Harris Hip Score is reliable and valid. The Harris hip score scale is composed of ten items and divided into four sub-scales: pain, function, absence of deformity, and range of motion. It is scored between 0 and 100 points. The criteria for evaluation are as follows: A score of less than 70 is considered poor, 70 to 80 is fair, 80 to 90 is good, and a score between 90 and 100 is excellent. To measure the range of motion sub-step of the Harris hip score, a universal goniometer was utilized in the investigation.
Length of hospital stay | 1-2 weeks
  The hospital stay was calculated from the patients hospitalized untill the discharged. The lenght of hospital was calculated as days.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahcesehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No